CLINICAL TRIAL: NCT00155532
Title: Skin Denervation in Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9261700704
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-06

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Peripheral neuropathy;systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

INTERVENTIONS:
Procedure: 3 mm-punch biopsies of the skin

SUMMARY:
To address the issues of skin denervation and its clinical and pathological correlations in systemic lupus erythematosus

DETAILED DESCRIPTION:
To address the issues of skin denervation and its clinical and pathological correlations in lupus, we will study a systemic lupus erythematosus (SLE) cohort by evaluating the extent of cutaneous innervation. Patients are recruited from the rheumatologic clinic, and various neuropsychiatric syndromes are diagnosed based on clinical judgement following detailed history taking and neurological examinations. Skin biopsy with PGP 9.5 immunohistochemistry will be performed following established procedures after informed consent is obtained, and punches of 3 mm in diameter will be taken from the lateral side of the distal leg, 10 cm above the lateral malleolus. Intraepidermal nerve fibre densities will be compared with results of immunological, pathological, psychophysical, and electrophysical studies to understand the pathogenesis of peripheral neuropathy in SLE.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of systemic lupus erythematosus based on the consensus criteria

Exclusion Criteria:

* Conditions known to be associated with peripheral neuropathy, such as diabetes, uremia, alcoholism, and the administration of potentially neurotoxic agents, such as alkylating agents, methotrexate, cyclosporine, and antibiotics.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-04; Study Completion 2004-03

PRIMARY OUTCOMES:
Quantitation of epidermal innervation

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Tsang Hsieh, MD, PhD, Study Director — Department of Neurology, National Taiwan University Hospital, 7 Chung-Shan S Rd., Taipei 100, Taiwan
Locations (1):
- Departments of Neurology, National Taiwan University Hospital, Taipei, Taiwan